CLINICAL TRIAL: NCT04203862
Title: A Phase 1 Single Ascending Dose Study of NPC-22 in Healthy Adult Males
Brief Title: A Study of NPC-22 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NPC-22
Record Dates: First submitted 2019-11-17; First posted 2019-12-18 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): Single administration of low dose NPC-22
  Interventions: Drug: NPC-22
- 2 (Experimental): Single administration of low/middle dose NPC-22
  Interventions: Drug: NPC-22
- 3 (Experimental): Single administration of middle dose NPC-22
  Interventions: Drug: NPC-22
- 4 (Experimental): Single administration of middle/high dose NPC-22
  Interventions: Drug: NPC-22
- 5 (Experimental): Single administration of high dose NPC-22
  Interventions: Drug: NPC-22
- 6 (Experimental): Single administration of placebo dose NPC-22
  Interventions: Drug: NPC-22 Placebo

INTERVENTIONS:
Drug: NPC-22 — Single administration of low dose NPC-22
  Arms: 1
Drug: NPC-22 — Single administration of low/middle dose NPC-22
  Arms: 2
Drug: NPC-22 — Single administration of middle dose NPC-22
  Arms: 3
Drug: NPC-22 — Single administration of middle/high dose NPC-22
  Arms: 4
Drug: NPC-22 — Single administration of high dose NPC-22
  Arms: 5
Drug: NPC-22 Placebo — Single administration of NPC-22 Placebo
  Arms: 6

SUMMARY:
The purpose of this trial is to examine the safety and pharmacokinetics of NPC-22 administered in a single ascending dose in healthy adult males.

DETAILED DESCRIPTION:
The healthy adult males will be randomized into six arms, and will receive single dose of NPC-22 (five doses, placebo)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have provided their own written informed consent
2. Subjects aged ≥20 and <40 years at the time of informed consent
3. Subjects with body weight of ≥50 kg and body mass index (BMI) (kg/m2) of ≥18.5 and <25.0
4. Subjects who were identified to have no health problem on physical examination, physical assessment, laboratory tests, or other examinations at screening by the principal investigator or a sub-investigator

Exclusion Criteria:

1. Subjects with a complication or a history of drug abuse (use of an illicit drug) or alcohol dependence
2. Subjects with a history of severe disease that may recur during the study period
3. Subjects with any concurrent illnesses
4. Subjects who received another study drug within 180 days prior to the start of study drug administration
5. Subjects who donated blood of ≥400 mL within 12 weeks, blood of ≥200 mL within 4 weeks, or blood components within 2 weeks prior to the start of the study
6. Subjects who used any medicinal product (including over the counter drugs except for topical products) or similar product like a dietary supplement (including health food) within 7 days prior to the start of study drug administration
7. Subjects who took any food or beverage containing grapefruit or St. John's wort within 7 days prior to the start of study drug administration
8. Subjects who took any alcohol or caffeine-containing beverage within 3 days prior to the start of study drug administration
9. Subjects who smoked within 90 days prior to the start of study drug administration, or do not agree to stop smoking during the study period
10. Subjects who had a positive result for HBs antigen, HCV antibody, or HIV antigen/antibody, or a positive reaction to syphilis serology or urine drug test at screening
11. Subjects who are unsuitable as a subject in this study in the judgement of the principal investigator or a sub-investigator based on the 12-lead electrocardiogram at screening [e.g., Fridericia's corrected QT (QTcF) interval of ≥450 ms]
12. Subjects who have a familial history of torsades de pointes or long QT syndrome
13. Subjects who are unsuitable as a subject in this study in the judgement of the principal investigator or a sub-investigator by having a deviation from the institutional reference values
14. Subjects who are unsuitable as a subject in this study in the judgement of the principal investigator or a sub-investigator due to other reasons

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Adverse events | 0-7 days post dose
  An adverse event will refer to any unfavorable or unintended sign (including an abnormal laboratory finding and abnormality on the 12-lead ECG or in vital signs) and symptom
Body temperature | 0-7 days post dose
  Body temperature will be measured for assess the safety of single ascending dose of NPC-22
Blood pressure | 0-7 days post dose
  Blood pressure will be measured for assess the safety of single ascending dose of NPC-22
Pulse rate | 0-7 days post dose
  Pulse rate will be measured for assess the safety of single ascending dose of NPC-22
ECG | 0-7 days post dose
  RR, PR, QRS, QT and QTcF interval and heart rate will be measured for assess the safety of single ascending dose of NPC-22
Number and/or rates of subjects with treatment-related adverse events as assessed by hematology tests | 0-7 days post dose
  Hematology tests will be performed for assessment the safety of single ascending dose of NPC-22
Number and/or rates of subjects with treatment-related adverse events as assessed by blood chemistry tests | 0-7 days post dose
  Blood chemistry tests will be performed for assessment the safety of single ascending dose of NPC-22
Number and/or rates of subjects with treatment-related adverse events as assessed by urinalysis | 0-7 days post dose
  Urinalysis will be performed for assessment the safety of single ascending dose of NPC-22

SECONDARY OUTCOMES:
Observed plasma concentration | 0-7 days post dose
Observed urine concentration | 0-4 days post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Shinanokai Shinanozaka Clinic, Shinjuku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided